CLINICAL TRIAL: NCT06135077
Title: Evaluation of Titanium-prepared Platelet-rich Fibrin in Bone Regeneration in Lateral Window Maxillary Sinus Augmentation (Clinical Trial)
Brief Title: Titanium Prepared Platelet-rich Fibrin in Bone Regeneration in Lateral Window Maxillary Sinus Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0301_10/2021
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Sinus Lifting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-PRF (Experimental)
  Interventions: Other: T-PRF alone
- T-PRF/xenograft (Active Comparator)
  Interventions: Other: T-PRF/Xenograft

INTERVENTIONS:
Other: T-PRF alone — T-PRF is the material to be tested in this study as an alternative to classical bone graft
  Arms: T-PRF
Other: T-PRF/Xenograft — One part of T-PRF will be divided into minute pieces to be mixed with xenograft
  Arms: T-PRF/xenograft

SUMMARY:
This trial aims to evaluate the effect of the sole use of T-PRF in bone formation process as applied in maxillary sinus floor elevation in comparison to traditional T-PRF/bone graft combination.

This study is clinical trial that will include 18 patients seeking implant placement in upper posterior maxilla compromised with maxillary sinus pneumatization. Patients will be assigned into control and test groups. All the patients will undergo sinus lifting procedure through which a combination of xenograft and T-PRF was used in the control group whereas; sole T-PRF will be applied in the test group.

ELIGIBILITY:
Inclusion Criteria:

* Systemically in a healthy condition.
* Residual bone height is ≤5mm in the posterior maxilla as measured with CBCT.
* Non-smokers.
* Good oral hygiene as indicated by plaque and bleeding scores

Exclusion Criteria:

* Medically compromised conditions will be excluded to avoid infections or any adverse reaction related to immunity suppression.
* Acute maxillary sinusitis.
* Patients administering any antibiotics or regular anti-inflammatory drugs.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Change in pain level | up to 2 weeks
  measuring level of pain using visual analog scale (VAS) 0-10, where 0 reading indicates no pain and 10 reading reflects the most severe pain.
Change in bone volume | up to 3 months
  pre opertaive and post operative CBCT
Change in bone denisty | up to 3 months
  pre opertaive and post operative CBCT
Change in bone height | up to 3 months
  pre opertaive and post operative CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt